CLINICAL TRIAL: NCT03554993
Title: A Phase I, Randomized, Single-center, 3-part Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Ascending Doses of CC 99677 in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Doses of CC-99677 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CC-99677-CP-001; U1111-1213-8860 (Other: WHO); 2017-004849-24 (EudraCT Number)
Record Dates: First submitted 2018-05-24; First posted 2018-06-13 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; Safety; CC-99677

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CC-99677 Under Fasted Conditions (Experimental): CC-99677 Under Fasted Conditions
  Interventions: Drug: CC-99677
- Placebo (Experimental): Placebo under fasted conditions
  Interventions: Other: Placebo
- CC-99677 Under Fed Conditions (Experimental): CC-99677 Under Fed Conditions
  Interventions: Drug: CC-99677

INTERVENTIONS:
Drug: CC-99677 — CC-99677
  Arms: CC-99677 Under Fasted Conditions; CC-99677 Under Fed Conditions
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a phase 1, randomized, single-center, 3-part, FIH study to assess the safety, tolerability, pharmacokinetics (PK, or how the drug behaves in the body), and pharmacodynamics (PD, or what the drug does to the body) of single and multiple doses of CC-99677 and to characterize the effect of food on the single-dose PK of CC-99677 in healthy adult subjects.

DETAILED DESCRIPTION:
This first-in-human (FIH) study aims to identify a safe and tolerable dose of CC 99677 in support of phase 2 and/or phase 3 studies to be conducted in subjects with underlying inflammatory diseases.

The study also aims to evaluate the PK of CC-99677 following administration of single and multiple oral doses, including assessment of the effect of food on the single dose PK of CC 99677, and to assess the effect of CC 99677 on electrocardiogram (ECG) parameters in healthy adult subjects. The pharmacodynamics (PD) and pharmacogenomics (PG) of CC 99677 will also be assessed.

Parts 1 and 2 are designed to evaluate the safety, tolerability, PK, and PD of single and multiple ascending doses of CC 99677, respectively. The study has been designed to allow for safety, tolerability, and PK data to be gathered in a stepwise fashion. Part 1 will consist of escalating single doses in sequential groups. Approximately 48 subjects will be enrolled into 6 planned dose level cohorts. Part 2 will consist of escalating multiple doses (administered for 14 days) in sequential groups. In Part 2, approximately 40 subjects will be enrolled into 5 proposed dose level cohorts. Each dose level cohort will consist of 8 subjects; 6 subjects will receive CC-99677 and 2 subjects will receive placebo according to the randomization schedule. In both Part 1 and Part 2, a higher daily dose level will not be initiated until adequate information on the preceding dose level is available and reviewed. Parts 1 and 2 will also employ strict dose escalation, individual subject, and intra cohort stopping criteria. Parts 1 and 2 will be placebo controlled to appropriately characterize the safety and tolerability of CC 99677.

Part 3 is designed to characterize the effect of food on the single dose PK of CC 99677.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is ≥ 18 and ≤ 55 years of age at the time of signing the informed consent form (ICF).
2. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Subject is in good health, as determined by the Investigator based on a physical examination at screening.
5. Female subjects of childbearing potential (FCBP) must:

   * Have 2 negative pregnancy tests as verified by the Investigator prior to the first dose of IP. She must agree to ongoing pregnancy testing during the course of the study, and prior to discharge from the study site. This applies even if the FCBP subject practices true abstinence from heterosexual contact.
   * Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis, as applicable, and source documented) or agree to use, and be able to comply with, one highly effective method and one effective barrier method of contraception without interruption, during the study (including any dose interruptions), and for at least 30 days after discontinuation of IP. The female subject's chosen form of highly effective contraception must be effective by the time the female subject is enrolled into the study (eg, hormonal contraception should be initiated at least 28 days prior to enrollment).
6. Female subjects NOT of childbearing potential must:

   - Have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation is required) at least 6 months before screening, or be postmenopausal (defined as 24 consecutive months without menses before screening, with a follicle-stimulating hormone [FSH] level of > 40 IU/L at screening).
7. Male subjects must:

   - Practice true abstinence (which must be reviewed on a monthly basis, as applicable, and source documented) or agree to use a condom during sexual contact with a pregnant female or a FCBP while participating in the study, during any dose interruptions, and for at least 90 days after discontinuation of IP, even if he has undergone a successful vasectomy. In addition, any non-pregnant FCBP partner of a male subject must use an approved method of effective contraception, without interruption, during the study (including any dose interruptions) and for at least 30 days after discontinuation of IP. Examples of approved methods of effective contraception for non-pregnant FCBP partners include progestogen-only oral hormonal contraception; male or female condom with or without spermicide; or cap, diaphragm, or sponge with spermicide.
8. Subject has a body mass index (BMI) ≥ 18 and ≤ 33 kg/m2 at screening.
9. Subject has clinical laboratory safety test results that are within normal limits or considered not clinically significant by the Investigator. In addition, ALT, AST, and total bilirubin must be ≤ the upper limit of normal at screening and on Day -1 (of Period 1, when applicable [ie, in Part 3]). Platelet count, absolute neutrophil count (ANC), and absolute lymphocyte count (ALC) must be ≥ the lower limit of normal at screening and on Day -1 (of Period 1, when applicable [ie, in Part 3]).
10. Subject is afebrile, with supine systolic blood pressure (BP) ≥ 90 and ≤ 140 mmHG, supine diastolic BP ≥ 50 and ≤ 90 mmHg, and pulse rate ≥ 40 and ≤ 110 bpm at screening.
11. Subject has normal or clinically acceptable 12-lead ECG. In addition:

    * If female, subject has a QTcF value ≤ 450 msec at screening.
    * If male, subject has a QTcF value ≤ 430 msec at screening.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any significant medical condition (including but not limited to neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, or other major disorders), laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Subject has any condition that confounds the ability to interpret data from the study.
4. Subject is pregnant or breastfeeding.
5. Subject was exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer).
6. Subject has used any prescribed systemic or topical medication (including but not limited to analgesics, anesthetics, etc) within 30 days prior to the first dose administration.

   Exceptions may apply on a case-by-case basis if considered not to interfere with the study objectives as agreed to by the Investigator and Sponsor's Medical Monitor.
7. Subject has used any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days prior to the first dose administration. Exceptions may apply on a case-by-case basis if considered not to interfere with the study objectives as agreed to by the Investigator and Sponsor's Medical Monitor.
8. Subject has used CYP3A inducers and/or inhibitors (including St. John's Wort) within 30 days preceding the first dose administration. The Indiana University (2016) "Cytochrome P450 Drug Interaction Table" should be utilized to determine inducers and/or inhibitors of CYP3A (http://medicine.iupui.edu/clinpharm/ddis/table.aspx). The Sponsor's Medical Monitor or designee should be queried in case of uncertainty.
9. Subject has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism, or excretion, eg, bariatric procedure. Appendectomy and cholecystectomy are acceptable. Other previous surgeries may be acceptable with concurrence of the Sponsor's Medical Monitor.
10. Subject donated blood or serum within 8 weeks before the first dose administration to a blood bank or blood donation center.
11. Subject has a history of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM; American Psychiatric Association, 2013]) within 2 years before the first dose administration, or positive drug screening test reflecting consumption of illicit drugs.
12. Subject has a history of alcohol abuse (as defined by the current version of the DSM [American Psychiatric Association, 2013]) within 2 years before the first dose administration, or positive alcohol screen.
13. Subject is known to have a history of hepatitis B and/or hepatitis C, or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at screening.

    Note: Subjects who received hepatitis B vaccination and who test positive for hepatitis B surface antibody and negative for both hepatitis B surface antigen and hepatitis B core antibody remain eligible for study participation.
14. Subject smokes > 10 cigarettes per day, or the equivalent in other tobacco products (self-reported).
15. Subject has received immunization with a live or live attenuated vaccine within 2 months prior to the first dose administration or is planning to receive immunization with a live or live attenuated vaccine for 2 months following the last dose administration.
16. Subject has a history of Gilbert's syndrome or has laboratory findings at screening that, in the opinion of the Investigator, are indicative of Gilbert's syndrome.
17. Subject has a history of incompletely treated Mycobacterium tuberculosis (TB) infection, as indicated by:

    * Subject's medical records documenting incomplete treatment for Mycobacterium TB.
    * Subject's self-reported history of incomplete treatment for Mycobacterium TB. Note: Subjects with a history of TB who have undergone treatment accepted by the local health authorities (documented) may be eligible for study entry.
18. Applicable to Part 2 only: subject has a positive QuantiFERON®-TB Gold (or equivalent) test at screening or 2 successive indeterminate QuantiFERON®-TB Gold (or equivalent) tests at screening.
19. Subject is part of the study site staff personnel or a family member of the study site staff.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | From enrollment until at least 28 days after completion of treatment
  Number of subjects with adverse events

SECONDARY OUTCOMES:
Pharmacokinetics - Cmax | up to 28 days
  Maximum observed plasma concentration
Pharmacokinetics - Tmax | up to 28 days
  Time to Cmax
Pharmacokinetics - AUC0-∞ | up to 28 days
  Area under the plasma concentration-time curve from time zero extrapolated to infinity
Pharmacokinetics - AUC0-t | up to 28 days
  Area under the plasma concentration-time curve from time zero extrapolated to the last quantifiable concentration
Pharmacokinetics - t1/2,z | up to 28 days
  Terminal elimination half-life
Pharmacokinetics - CL/F | up to 28 days
  Apparent total clearance
Pharmacokinetics - Vz/F | up to 28 days
  Apparent total volume of distribution
Effect of CC-99677 on electrocardiogram (ECG) parameters | up to 24 hours after single dose administration
  ECG data will be collected using continuous 12 lead digital Holter recorders at prespecified timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Ramirez-Valle, MD, PhD, Study Director — Celgene
Locations (1):
- Quotient Clinical, Ruddington, United Kingdom

REFERENCES:
- [Derived] Gaur R, Mensah KA, Stricker J, Adams M, Parton A, Cedzik D, Connarn J, Thomas M, Horan G, Schafer P, Mair S, Palmisano M, Ramirez-Valle F. CC-99677, a novel, oral, selective covalent MK2 inhibitor, sustainably reduces pro-inflammatory cytokine production. Arthritis Res Ther. 2022 Aug 18;24(1):199. doi: 10.1186/s13075-022-02850-6. PMID 35982464
- [Derived] Malona J, Chuaqui C, Seletsky BM, Beebe L, Cantin S, Kalken DV, Fahnoe K, Wang Z, Browning B, Szabo H, Koopman LA, Oravecz T, McDonald JJ, Ramirez-Valle F, Gaur R, Mensah KA, Thomas M, Connarn JN, Hu H, Alexander MD, Corin AF. Discovery of CC-99677, a selective targeted covalent MAPKAPK2 (MK2) inhibitor for autoimmune disorders. Transl Res. 2022 Nov;249:49-73. doi: 10.1016/j.trsl.2022.06.005. Epub 2022 Jun 9. PMID 35691544